CLINICAL TRIAL: NCT01039974
Title: An Open-label, Randomized, Single Sequence, Two Period Study to Assess the Effect of Repeat Oral Dosing of Ketoconazole on the Pharmacokinetics of a Single Oral Dose of GSK962040 in Healthy Volunteers
Brief Title: GSK962040 Drug-drug Interaction Study With Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112648
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Gastroparesis
Keywords: ketoconazole; GSK962040; Drug-Drug Interaction; Phase I
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohorts 1-2 (Experimental): Cohorts 1 and 2 will complete both periods Period 1 GSK962040 single dose Period 2 Ketoconazole repeat dose (10 days), GSK962040 single dose
  Interventions: Drug: GSK962040; Drug: Ketoconazole

INTERVENTIONS:
Drug: GSK962040 — GSK962040. Planned doses per cohort as follows:
  Cohort 1 planned dose = 10 mg; Cohort 2 to be determined based on data from Cohort 1
Drug: Ketoconazole — 400 mg

SUMMARY:
This study will determine the effect of 400 mg ketoconazole on the pharmacokinetics of a single dose of GSK962040. The results from this study will help to estimate the maximum increase in exposure during concomitant use of strong CYP3A4 inhibitors. This study will also contain an exploratory investigation of biliary secretion of GSK962040 and or its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. In any case, liver function tests must be strictly within the normal range at screening.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory].
* Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for at least 5 days following the last dose of study medication. GSK962040 and ketoconazole are defined as study medications.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication through at least 5 days following the last dose of study medication. GSK962040 and ketoconazole are defined as study medications.
* Body weight > or = 50 kg and BMI within the range 18.5-29.9 kg/m2 (inclusive).
* Capable of giving written informed consent
* QTcB or QTcF < 450 msec or QTc<480msec in subjects with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period.
* Normal physical examination (physical exam demonstrates no evidence of clinically active disease or physical or mental impairment). A subject with a clinical abnormality may be included only if the Principal Investigator or physician designee considers that the abnormality will not introduce additional risk factors and will not interfere with the study procedures. Consultation with the GSK medical monitor is required before such subjects may be included.

Exclusion Criteria:

* History of major gastrointestinal surgical procedure.
* History of cholecystectomy or biliary tract disease.
* A history or presence of recreational drug abuse or dependence or current abuse as evidenced by positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test (from the first urine of the day) at screening or prior to dosing.
* Lactating or pregnant females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09-18 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (AUC(0-inf), and Cmax) of GSK962040 | Duration of dosing

SECONDARY OUTCOMES:
Safety and tolerability assessments, consisting of AEs, ECGs, vital signs, clinical laboratory tests. | Duration of dosing
Additional pharmacokinetic parameters of GSK962040, i.e., tmax, t1/2, AUC(0-t) | Duration of dosing
To characterize the nature of the GSK962040-related material in plasma, 24-hour urine, and bile. | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112648 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112648?search=study&search_terms=112648#rs
- Available data/document: Annotated Case Report Form: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register